CLINICAL TRIAL: NCT07234383
Title: Accelerated HEmodiafiltration in Severe Acute Diquat (AHEAD) Poisoning: a Single-center, Single-arm, Open-label, Clinical Trial
Brief Title: Accelerated HEmodiafiltration in Severe Acute Diquat (AHEAD) Poisoning
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hao Sun, Principal Investigator, Clinical Associate Professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0919-1
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Diquat Poisoning
MeSH Terms: interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Accelerated Initiation (Experimental): Participants in this experimental arm will receive CVVHDF within 12 hours of eligibility confirmation. This 12-hour window includes the time required to obtain consent, place a dialysis catheter, and initiate CVVHDF.
  Interventions: Procedure: Continuous Veno-Venous Hemodiafiltration

INTERVENTIONS:
Procedure: Continuous Veno-Venous Hemodiafiltration — CVVHDF will be delivered following hemoperfusion with a dialysate-to-replacement fluid ratio maintained at 1:1, a blood flow rate of 150-200 mL/min, and a target dialysis dose of 30 mL/kg/h (excluding additional fluid removal). Regional anticoagulation (e.g., heparin or other agent per device requirements) will be used to prevent clotting within the circuit. Once CVVHDF is initiated in either arm, it will not be discontinued until one of the following encountered: (i) death; or (ii) a change in goals of care with withdrawal of life-sustaining interventions; or (3) recovery of kidney function, as determined by treating clinician(s), such that CVVHDF will be no longer required. However, CVVHDF will be reinitiated at the discretion of treating clinician(s), if kidney function comes suboptimal after a period of discontinuation.

SUMMARY:
Diquat (1,1'-ethylene-2,2'-bipyridinium) is a bipyridine herbicide that shares a similar physicochemical structure and redox cycling mechanism with paraquat. Upon ingestion, it is rapidly absorbed and distributes widely, including gastrointestinal tract, kidneys, liver, skeletal muscle, lungs, myocardium, and central nervous system. Severe diquat poisoning commonly causes toxic encephalopathy, circulatory collapse, and multiorgan dysfunction. Extracorporeal treatments, including hemoperfusion, hemodialysis, and continuous kidney replacement therapy, are frequently used in management. Continuous veno-venous hemodiafiltration (CVVHDF), the most frequently used continuous kidney replacement therapy modality, is primarily indicated for acute kidney injury. Acute kidney injury occurs in up to 73.3% of patients with acute diquat poisoning, and nearly all patients with severe acute diquat poisoning are at risk of developing acute kidney injury. In clinical practice, patients with severe acute diquat poisoning are typically defined as those with a plasma diquat concentration of ≥1000 ng/mL measured at the time of presentation to the emergency department. However, the Extracorporeal Treatments in Poisoning (EXTRIP) workgroup has not issued any definitive recommendations on initiating extracorporeal treatments for diquat poisoning, and the optimal timing for starting CVVHDF has not been evaluated in clinical trials. Current practice typically delays CVVHDF until acute kidney injury occurs. A preliminary retrospective cohort study suggested that, among severe acute diquat poisoning patients treated with combined hemoperfusion and CVVHDF, an interval of <30 minutes between hemoperfusion and CVVHDF was associated with a significantly lower risk of death compared with longer intervals (≥30 minutes). Accordingly, this study proposes a single-arm trial (SAT) to determine whether accelerated initiation of CVVHDF immediately following hemoperfusion improves outcomes in patients with severe acute diquat poisoning.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥ 18 years; and
2. A history of oral exposure to diquat solution, reported by patient(s) or their legal proxies; and
3. An exposure time (time form exposure to presentation at ED) ≤ 48 hours, reported by patient(s) or their legal proxies; and
4. Plasma diquat concentration measured upon ED presentation ≥ 1,000 ng/mL.

Exclusion criteria:

1. Evidence of co-ingestion of other toxic substances alongside diquat; and/or
2. Withholding of CVVHDF due to limitations on the escalation of life-sustaining therapies; and/or
3. Any CKRT within the previous 2 months; and/or
4. Kidney transplant within the past 365 days; and/or
5. Known pre-hospitalization advanced chronic kidney disease, defined by an estimated glomerular filtration rate calculated using serum creatine (eGFRer) of less than 30 mL/min/1.73 m2 by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation, if pre-hospitalization serum creatine is available; and/or (6) Treating clinician(s) believe(s) that either immediate or deferral of CVVHDF initiation is mandated; and/or (7) Pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality rate | 90 days within the index date of randomization
Time from exposure to death | 90 days within the index date of randomization
  The primary outcome measure included time from exposure to death.

SECONDARY OUTCOMES:
ICU-free days | 90 days within the index date of randomization
Ventilator-free days | 90 days within the index date of randomization
Vasoactive-free days | 90 days within the index date of randomization
CVVHDF dependence rate | 90 days within the index date of randomization
Hospitalization-free days | 90 days within the index date of randomization
Major adverse kidney events rate | 90 days within the index date of randomization
  The secondary outcome measure included major adverse kidney events at 90 days after randomization, defined as the composite of death, CVVHDF dependence, or sustained reduction of kidney function (defined as eGFR <75% of the lowest eGFR measured during hospitalization).